CLINICAL TRIAL: NCT05681039
Title: Phase 2 Trial of Neoadjuvant and Adjuvant Tiragolumab Plus Atezolizumab in Patients With Newly Diagnosed PD-L1 CPS Positive Resectable Stage 3-4 Oral Cavity Squamous Cell Carcinoma (OCSCC).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0446; NCI-2022-10637 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Tiragolumab; atezolizumab; Standard of Care; Surveys and Questionnaires; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant and Adjuvant (Experimental)
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Behavioral: Standard of Care; Behavioral: Questionnaires; Radiation: Cisplatin; Radiation: Carboplatin

INTERVENTIONS:
Drug: Tiragolumab — Given by IV (vein)
Drug: Atezolizumab — Given by IV (vein)
  Other Names: MPDL3280A; TECENTRIQ
Behavioral: Standard of Care — after care from surgery
Behavioral: Questionnaires — Quality of life
Radiation: Cisplatin — Given by IV (vein)
Radiation: Carboplatin — Given by IV (vein)

SUMMARY:
To learn if treatment with tiragolumab and atezolizumab before and after standard of care surgery and chemoradiation (radiation therapy with or without cisplatin/carboplatin) can help to control OCSCC that is PD-L1 CPS positive.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the major pathological response rate, defined as <10% viable tumor in the resection specimen, after two cycles of neoadjuvant atezolizumab and tiragolumab in patients with newly diagnosed, local-regionally advanced OCSCC that is PD-L1 CPS ≥1. Response at the primary site and in nodal disease will be evaluated.

Secondary Objectives:

To evaluate the safety of two cycles of atezolizumab and tiragolumab in patients with newly diagnosed, local-regionally advanced OCSCC, as measured by the incidence, nature and severity of adverse events with severity measured by CTCAE V5.

To evaluate the overall response rate (ORR) as measured by RECIST1.1 after two cycles of neoadjuvant atezolizumab and tiragolumab, including complete or partial response (CR+PR).

To evaluate the distribution of percent tumor viability in tumor biopsies and resection specimens after two cycles of atezolizumab and tiragolumab.

To estimate the 12, 18 and 24 month progression-free survival (PFS, defined as time from enrollment to date of progression or death) and overall survival (OS, defined as time from enrollment to death) in the study population.

Exploratory Objectives:

To investigate changes in the tumor microenvionment before and after two cycles of atezolizumab and tiragolumab as measured by multispectral immunofluorescence and single-cell sequencing.

To genetically profile OSCC by use of oral rinse and to measure changes in patient-specific somatic mutations by cfDNA before, during and after neoadjuvant immunotherapy.

To assess polyfunctionality in peripheral blood CD4+ and CD8+ T cells after neoadjuvant immunotherapy, radiotherapy and adjuvant immunotherapy.

To evaluate the symptom severity mean (measured by MDASI-HN), and its association with the major pathological response.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age 18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically confirmed, newly diagnosed, OCSCC that is clinical AJCC 8th edition Stage 3-4 (T1-T4N1-3, T3-T4N0)
* Patients with a history of previously resected stage T1N0 or T2N0 OCSCC and no prior history of radiotherapy to the head and neck are eligible at local +/- regional recurrence if they otherwise meet stage criteria.
* Surgically resectable OCSCC as determined by the patients' treating head and neck surgeon. Patients with a clinical diagnosis of oral cavity cancer, awaiting a biopsy are eligible to consent for pre-screening.
* Measurable disease per RECIST v1.1
* PD-L1 CPS≥ 1 (determined by immunohistochemistry with the 22C3 antibody) as documented through testing of a representative tumor tissue specimen
* Availability of a representative tumor specimen for exploratory biomarker research (see Appendix 12 for information on tumor specimens) A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 15 slides containing unstained, freshly cut, serial sections must be available for baseline biomarker analysis along with an associated pathology report prior to study enrollment. If archival tumor tissue is unavailable or is determined to be unsuitable for, tumor tissue must be obtained from a biopsy performed at screening.
* ECOG Performance Status of 0-1
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * ANC 1.5 109/L (1500/L) without granulocyte colony-stimulating factor support
  * Lymphocyte count 0.5 109/L (500/L)
  * Platelet count 100 109/L (100,000/L) without transfusion
  * Hemoglobin 90 g/L (9 g/dL) Patients may be transfused to meet this criterion.
  * AST, ALT, and alkaline phosphatase (ALP) 2.5 upper limit of normal (ULN)
  * Serum bilirubin 1.5 ULN with the following exception:

Patients with known Gilbert disease: serum bilirubin 3 ULN

* Creatinine clearance 50 mL/min (calculated using the Cockcroft-Gault formula)
* Serum albumin 25 g/L (2.5 g/dL)
* For patients not receiving therapeutic anticoagulation: INR and aPTT 1.5 xULN

  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
  * Negative HIV test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy for ≥3 months, have a CD4 count 200/µL, and have an undetectable viral load
  * Negative hepatitis B surface antigen (HBsAg) test at screening
  * Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:
* Negative total hepatitis B core antibody (HBcAb)
* Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL The HBV DNA test will be performed only for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.

  * Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
  * Requirements for contraception and pregnancy testing for a clinical trial should encompass all investigational medicinal products (IMPs) as well as protocol-mandated non-investigational medicinal products (NIMPs) such as background therapy, and the measures to be followed should be based on the medicinal product with the highest risk (see the protocol synopsis for definition of IMP and NIMP). Contraception requirements for marketed Genentech IMPs or NIMPs should be based on recommendations in the Summary of Product Characteristics (SmPC) or, if there is no SmPC, national prescribing information. Contraception requirements for unapproved Genentech IMPs or NIMPs should be based on recommendations in the Investigator Brochure (IB).
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

Women must remain abstinent or use contraceptive methods with a failure rate of 1% per year during the treatment period and for 5 months after the final dose of atezolizumab, 90 days after the last dose of tiragolimab and for 6 months after the final dose of carboplatin or cisplatin. Women must refrain from donating eggs during this same period.

A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state ( 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.

Examples of contraceptive methods with a failure rate of 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

- For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of 1% per year during the treatment period, for 90 days (a sperm cycle) after the final dose of tiragolumab and for 6 months after the final dose of carboplatin or cisplatin. Men must refrain from donating sperm during this same period.

With a pregnant female partner, men must remain abstinent or use a condom during the treatment period, for 90 days after the final dose of tiragolumab and for 6 months after the final dose of carboplatin or cisplatin to avoid exposing the embryo.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

* Positive test for SARS-CoV-2 within two weeks of enrollment.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium 1.5 mmol/L, calcium 12 mg/dL or corrected serum calcium ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 6 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.

Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

* Rash must cover 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months

  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
  * Active tuberculosis
  * Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
  * Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
  * History of malignancy within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
  * Severe infection, including SARS-CoV-2 infection, within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact patient safety.
  * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
  * Prior allogeneic stem cell or solid organ transplantation
  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
  * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study, or within 90 days after the final dose of tiragolumab or 5 months after the final dose of atezolizumab Patients being treated with chemotherapy (i.e., carboplatin and cisplatin) should not receive live vaccines.
  * Current treatment with anti-viral therapy for HBV
  * Positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening An EBV PCR test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
  * Prior treatment for head and neck cancer that includes in filed radiotherapy
  * Treatment with investigational therapy within 42 days prior to initiation of study treatment
  * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including antiCTLA-4, anti PD-1, and anti PD-L1 therapeutic antibodies
  * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
  * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antiTNF- agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.

Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

Patients may receive corticosteroids as anti-emetics during adjuvant (chemo)radiotherapy per the standard of care.

* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the chemotherapy regimen the patient may receive during the study.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The major pathological response rate after neoadjuvant atezolizumab and tiragolumab. | through study completion; an average of 1 year.
  To determine the major pathological response rate, defined as <10% viable tumor in the resection specimen, after two cycles of neoadjuvant atezolizumab and tiragolumab in patients with newly diagnosed, local-regionally advanced OCSCC that is PD-L1 CPS ≥1. Response at the primary site and in nodal disease will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wotman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org